CLINICAL TRIAL: NCT01000285
Title: Phase I/II Trial of Dose-Adjusted EPOCH Chemotherapy With Bortezomib Combined With Integrase Inhibitor Therapy for HTLV-1 Associated T-Cell Leukemia Lymphoma
Brief Title: EPOCH Chemotherapy and Bortezomib for Associated T-Cell Leukemia Lymphoma
Acronym: ATLL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-1758 / 201108212
Record Dates: First submitted 2009-10-19; First posted 2009-10-23 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Leukemia-Lymphoma, Adult T-Cell
MeSH Terms: conditions — Leukemia-Lymphoma, Adult T-Cell | interventions — Bortezomib; Etoposide; etoposide phosphate; Vincristine; Doxorubicin; Prednisone; Cyclophosphamide; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Bortezomib 1.0 mg/m2 intravenous (IV) Days 1-4
  Etoposide 50 mg/m2/d 96 hour continuous intravenous infusion (CIVI) on Days 1-4
  Vincristine 0.4 mg/m2/d 96 hour CIVI on Days 1-4
  Doxorubicin 10 mg/m2/d 96 hour CIVI on Days 1-4
  Prednisone 60 mg/m2/d PO on Days 1-5
  Cyclophosphamide 375 mg/m2 IV on Day 5
  Raltegravir 400 mg PO twice per day (BID) every day starting with cycle 2 therapy for the entire duration of the cycle.
  Cycles will be repeated every 21-28 days for 2 cycles beyond best response, or a maximum of 6 cycles.
  Interventions: Drug: Bortezomib; Drug: Etoposide; Drug: Vincristine; Drug: Doxorubicin; Drug: Prednisone; Drug: Cyclophosphamide; Drug: Raltegravir

INTERVENTIONS:
Drug: Bortezomib
  Other Names: Velcade®
Drug: Etoposide
  Other Names: Toposar®, VePesid®, Etopophos®
Drug: Vincristine
  Other Names: Oncovin ®, Vincasar Pfs ®
Drug: Doxorubicin
  Other Names: Adriamycin ®, Rubex ®
Drug: Prednisone
  Other Names: Deltasone®, Liquid Pred®, Meticorten®, Orasone®
Drug: Cyclophosphamide
  Other Names: Cytoxan ®, Neosar ®
Drug: Raltegravir
  Other Names: Isentress®

SUMMARY:
The rationale of the current study is to explore the use of combination chemotherapy together with antiretroviral agents in order to determine the efficacy and toxicity of this approach, while also examining markers of virus replication and expression, and tumor cell proliferation to gain understanding of the biological basis of this malignancy and to identify predictors of response.

DETAILED DESCRIPTION:
Primary Endpoint:

- To determine the tolerability and efficacy (response rate) of dose adjusted bortezomib-EPOCH (DA B-EPOCH) chemotherapy combined with Raltegravir in patients with HTLV-1 associated leukemia/lymphoma (ATLL).

Secondary Endpoints:

* To evaluate the effects of DA B-EPOCH chemotherapy combined with Raltegravir on HTLV-1 DNA and RNA load, HTLV-1 integrase gene sequence, and HTLV-1 integration sites. To determine if relapsed or progressive disease is a result of renewed virus replication.
* To evaluate the relation of NFκB gene expression profile on response to DA B-EPOCH chemotherapy combined with Raltegravir.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented ATLL. Patients with previously untreated or treated ATLL are eligible.
* Tumors must be CD3 positive (>50% cells express CD3).
* Documented HTLV-1 infection: documentation may be serologic assay (ELISA, Western blot) Confirmation of HTLV-1 rather than HTLV-2 by differential Western blot (e.g. Genelabs Diagnostics HTLV Blot 2.4) or PCR is desirable but his result is not required prior to trial enrollment.
* Measurable disease must be present. These nodes or masses should be selected according to all of the following: they should be clearly measurable in at least two perpendicular dimensions; if possible they should be from disparate regions of the body; and they should include mediastinal and retroperitoneal areas of disease whenever these sites are involved.For patients with acute (leukemic) form of ATLL, measureable disease can be derived from CD4+ lymphocyte flow data on the peripheral blood and/or bone marrow.
* All stages are eligible.
* Adequate hematologic function within 14 days before enrollment: ANC>1000 cells/mm3, platelet count>75,000 cells/mm3 unless cytopenias are secondary to ATLL. All patients must be off hematologic growth factors for at least 24 hrs.
* Adequate hepatic function, transaminase <3 times the upper limit of normal unless due to to Gilbert's disease or hepatic involvement by tumor; total bilirubin ≤1.5 times the upper limit of normal
* Creatinine<2.0 unless due to lymphoma.
* Karnofsky Performance Status (KPS) at least 50
* Age at least 18. -Voluntary written informed consent before performance of any study- related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female patients of child bearing potential must have a negative pregnancy test within 72 hrs of initiation of therapy. Female patients are either post-menopausal or surgically sterilized or willing to use two acceptable methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) during the study. Male patients must agree to use two acceptable methods for contraception for the duration of the study. Women must avoid pregnancy and men avoid fathering children while in the study.
* HIV positive patients are eligible if they are receiving at least two other active anti-HIV therapies other than zidovudine or atazanavir.
* Patients with active hepatitis B (HBV) infection are eligible if they are receiving effective anti-HBV therapy.
* Inclusion of Women and Minorities: Both men and women and members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Acute active infection requiring acute therapy. Chronic therapy with potentially myelosuppressive agents is allowed provided that entry hematologic criteria are met.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Women who are pregnant or breastfeeding. Confirmation that the subject is not pregnant must be established by a negative serum B-human chorionic gonadotropin (B-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has ≥Grade 2 peripheral neuropathy
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any electrocardiogram (ECG) abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

  * 1.5x upper limit of normal (ULN) total bilirubin except if is determined to be related to Gilbert's disease or tumor biliary/liver involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-09; Primary Completion 2014-05 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ratner, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (6):
- United States (6):
  - University of Miami Hospital/Sylvester, Miami, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University, College of Physicians and Surgeons, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- [Background] Ratner L, Harrington W, Feng X, Grant C, Jacobson S, Noy A, Sparano J, Lee J, Ambinder R, Campbell N, Lairmore M; AIDS Malignancy Consortium. Human T cell leukemia virus reactivation with progression of adult T-cell leukemia-lymphoma. PLoS One. 2009;4(2):e4420. doi: 10.1371/journal.pone.0004420. Epub 2009 Feb 10. PMID 19204798
- [Background] Satou Y, Nosaka K, Koya Y, Yasunaga JI, Toyokuni S, Matsuoka M. Proteasome inhibitor, bortezomib, potently inhibits the growth of adult T-cell leukemia cells both in vivo and in vitro. Leukemia. 2004 Aug;18(8):1357-63. doi: 10.1038/sj.leu.2403400. PMID 15190257
- [Background] Mitra-Kaushik S, Harding JC, Hess JL, Ratner L. Effects of the proteasome inhibitor PS-341 on tumor growth in HTLV-1 Tax transgenic mice and Tax tumor transplants. Blood. 2004 Aug 1;104(3):802-9. doi: 10.1182/blood-2003-11-3967. Epub 2004 Apr 15. PMID 15090453
- [Background] Tsukasaki K, Hermine O, Bazarbachi A, Ratner L, Ramos JC, Harrington W Jr, O'Mahony D, Janik JE, Bittencourt AL, Taylor GP, Yamaguchi K, Utsunomiya A, Tobinai K, Watanabe T. Definition, prognostic factors, treatment, and response criteria of adult T-cell leukemia-lymphoma: a proposal from an international consensus meeting. J Clin Oncol. 2009 Jan 20;27(3):453-9. doi: 10.1200/JCO.2008.18.2428. Epub 2008 Dec 8. PMID 19064971
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 12/22/2010 and closed to participant enrollment on 05/29/2014.
Groups:
- EPOCH Chemotherapy & Bortezomib: Bortezomib 1.0 mg/m2 IV Days 1-4
  Etoposide 50 mg/m2/d 96 hour CIVI on Days 1-4
  Vincristine 0.4 mg/m2/d 96 hour CIVI on Days 1-4
  Doxorubicin 10 mg/m2/d 96 hour CIVI on Days 1-4
  Prednisone 60 mg/m2/d PO on Days 1-5
  Cyclophosphamide 375 mg/m2 IV on Day 5
  Raltegravir 400 mg PO BID every day starting with cycle 2 therapy for the entire duration of the cycle.
  Cycles will be repeated every 21-28 days for 2 cycles beyond best response, or a maximum of 6 cycles.
Period: Overall Study
Arm/Group | EPOCH Chemotherapy & Bortezomib
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Acute ATLL; Lymphoma ATLL: Bortezomib 1.0 mg/m2 IV Days 1-4
  Etoposide 50 mg/m2/d 96 hour CIVI on Days 1-4
  Vincristine 0.4 mg/m2/d 96 hour CIVI on Days 1-4
  Doxorubicin 10 mg/m2/d 96 hour CIVI on Days 1-4
  Prednisone 60 mg/m2/d PO on Days 1-5
  Cyclophosphamide 375 mg/m2 IV on Day 5
  Raltegravir 400 mg PO BID every day starting with cycle 2 therapy for the entire duration of the cycle.
  Cycles will be repeated every 21-28 days for 2 cycles beyond best response, or a maximum of 6 cycles.
- Total: Total of all reporting groups
Arm/Group | Acute ATLL | Lymphoma ATLL | Total
Number analyzed (Participants) | 6 | 12 | 18
Age, Continuous [Median (Full Range); unit: years] | 51.5 [38 to 70] | 56 [36 to 76] | 52 [36 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 14
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 6 | 12 | 18
Birthplace [Number; unit: participants]
  Antigua | 0 | 1 | 1
  Dominican Republic | 1 | 0 | 1
  Haiti | 0 | 3 | 3
  Jamaica | 3 | 5 | 8
  USA | 1 | 2 | 3
  Virgin Islands | 0 | 1 | 1
  Bahamas | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Treatment as Measured by Number of Participants With Grade 3 or Higher Adverse Events
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized for all toxicity reporting.
Time Frame: Up to 30 days after completion of treatment
Measure: Number; unit: participants
Arm/Group | EPOCH Chemotherapy & Bortezomib
Number analyzed (Participants) | 18
participants
  Fatigue | 1
  Vomiting | 1
  Spontaneous bacterial peritonitis | 1
  Abdominal distension | 2
  Hemoglobin | 6
  Leukocytes (WBC) | 7
  Lymphopenia | 1
  Neutrophils | 6
  Platelets | 6
  Infection without neutropenia | 1
  Infection with neutropenia | 1
  Omaya port infection | 1
  IV port infection | 1
  Sepsis | 2
  Neutropenic fever | 3
  Hypoglycemia | 1
  Hyperglycemia | 2
  Magnesium | 1
  Hypokalemia | 1
  Hypertriglyceridemia | 1
  Confusion | 1
  Headache | 1
  Encephalitis | 1
  Abdominal pain | 1
  Cough | 1
  Dyspnea | 1

2. Primary Outcome: Efficacy of Treatment as Measured by Best Overall Response
Description: -The response definitions used for this study are the 2007 Cheson criteria.
Time Frame: Up to 4 years following completion of therapy
Measure: Number; unit: participants
Arm/Group | EPOCH Chemotherapy & Bortezomib
Number analyzed (Participants) | 18
participants
  Progressive Disease | 3
  Stable disease | 3
  Partial response | 9
  Complete response | 3

3. Secondary Outcome: Time to Progression
Description: -The progression definitions used for this study are from the 2007 Cheson criteria.
Time Frame: Up to 4 years following completion of therapy
Population: 12 out of the 18 participants had a complete or partial response.
Measure: Median (Full Range); unit: days
Arm/Group | EPOCH Chemotherapy & Bortezomib
Number analyzed (Participants) | 18
days
  Best response of complete response | 199 [190 to 864]
  Best response of partial response | 143 [85 to 240]
  Best response of stable disease | 88 [55 to 116]
  All participants | 127 [23 to 864]

4. Secondary Outcome: Effects of on HTLV-1 DNA After Treatment as Measured by Proviral Loads
Time Frame: 6 months
Measure: Mean (Standard Error); unit: copies/peripheral blood mononuclear cell
Groups:
- Responders: Patients who had a complete or partial response to treatment
- Non-responders: Patients who had stable or progressive disease after treatment.
Arm/Group | Responders | Non-responders
Number analyzed (Participants) | 12 | 6
copies/peripheral blood mononuclear cell
  Baseline | 0.372 (0.123) | 0.417 (0.045)
  Study completion | 0.0128 (0.023) | 0.033 (0.147)

5. Secondary Outcome: Relation of NFκB Gene Expression Profile on Response
Description: Standard error represents the standard error of the fold expression of protein coding transcripts for each gene indicated.
Time Frame: 6 months
Population: Average RPKM values normalized to Patient A before therapy.
Measure: Mean (Standard Error); unit: fold expression
Arm/Group | Patient A (Responder) Pre-Therapy | Patient A (Responder) Post-Therapy | Patient B (Responder) Pre-Therapy | Patient B (Responder) Post-Therapy | Patient C (Non-responder) Pre-Therapy | Patient C (Non-responder) Post-Therapy | Patient D (Non-responder) Pre-Therapy | Patient D (Non-responder) Post-Therapy
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
fold expression
  BLK | 1.000 (0.000) | 0.178 (0.015) | 0.889 (0.150) | 0.172 (0.073) | 68.856 (10.543) | 77.590 (12.715) | 233.179 (60.619) | 46.801 (13.193)
  CADMI | 1.000 (0.000) | 0.011 (0.001) | 0.623 (0.031) | 0.007 (0.001) | 1.494 (0.190) | 1.816 (0.105) | 2.013 (0.085) | 0.470 (0.026)
  CD25 | 1.000 (0.000) | 0.035 (0.006) | 0.303 (0.013) | 0.015 (0.003) | 0.862 (0.013) | 0.691 (0.013) | 2.897 (0.098) | 0.512 (0.023)
  CD4 | 1.000 (0.000) | 1.380 (0.047) | 1.437 (0.080) | 0.607 (0.023) | 1.319 (0.075) | 1.923 (0.092) | 3.057 (0.340) | 0.648 (0.056)
  CD45 | 1.000 (0.000) | 1.718 (0.045) | 2.049 (0.035) | 0.959 (0.016) | 1.163 (0.021) | 1.640 (0.039) | 0.594 (0.008) | 0.714 (0.019)

6. Secondary Outcome: Effects of HTLV-1 RNA Load After Treatment as Measured by Hbz Messenger RNA
Time Frame: 6 months
Measure: Mean (Standard Error); unit: copies/peripheral blood mononuclear cell
Arm/Group | Responders | Non-responders
Number analyzed (Participants) | 12 | 6
copies/peripheral blood mononuclear cell
  Baseline | 37.0 (11.9) | 41.9 (29.1)
  Study completion | 7.33 (2.76) | 35.7 (23.7)

7. Secondary Outcome: Effects of HTLV-1 Integrase Gene Sequence After Treatment as Measured by Nucleotide Divergence
Time Frame: 6 months
Measure: Mean (Standard Error); unit: percentage of nucleotide divergence
Arm/Group | EPOCH Chemotherapy & Bortezomib
Number analyzed (Participants) | 18
percentage of nucleotide divergence
  Baseline | 0.49 (0.05)
  Study completion | 0.52 (0.06)

8. Secondary Outcome: Effects of HTLV-1 Integration Sites After Treatment
Time Frame: 6 months
Measure: Mean (Standard Error); unit: number of integration sites
Arm/Group | EPOCH Chemotherapy & Bortezomib
Number analyzed (Participants) | 18
number of integration sites
  Baseline | 1.31 (0.31)
  Study completion | 1.00 (0.22)

ADVERSE EVENTS:
Arm/Group | EPOCH Chemotherapy & Bortezomib
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EPOCH Chemotherapy & Bortezomib (N=18)
Sepsis (Infections and infestations) | 1 (18)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EPOCH Chemotherapy & Bortezomib (N=18)
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Albumin (Metabolism and nutrition disorders) | 4
Alkaline phosphtase (Investigations) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blurred vision (Eye disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Chills (General disorders) | 1
Confusion (Psychiatric disorders) | 2
Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Creatinine (Renal and urinary disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Dry eyes (Eye disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema (General disorders) | 2
Encephaltis (Infections and infestations) | 1
Extremity pain (Musculoskeletal and connective tissue disorders) | 1
Fatigue (General disorders) | 8
Fever (General disorders) | 2
GI bleed/ulcers (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 11
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 2
IV port infection (Infections and infestations) | 1
Indigestion (Gastrointestinal disorders) | 2
Infection with neutropenia (Infections and infestations) | 1
Infection without neutropenia (Infections and infestations) | 2
Leukocytes (WBC) (Investigations) | 8
Lymphopenia (Investigations) | 1
Magnesium (Metabolism and nutrition disorders) | 3
Mucositis (Gastrointestinal disorders) | 3
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Neutropenic fever (Infections and infestations) | 3
Neutrophils (ANC) (Investigations) | 7
Omaya port infection (Infections and infestations) | 1
Opthalmoplegia/laryngeal/aphasia (Nervous system disorders) | 1
Pigment changes (Skin and subcutaneous tissue disorders) | 1
Platelets (Investigations) | 8
Rash (Skin and subcutaneous tissue disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
SGOT (AST) (Investigations) | 4
SGPT (ALT) (Investigations) | 4
Seizure (Nervous system disorders) | 1
Sensory neuropathy (Nervous system disorders) | 9
Sepsis (Infections and infestations) | 1
Septic arthritis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Spontaneous bacterial peritonitis (Gastrointestinal disorders) | 1
Uric acid (Metabolism and nutrition disorders) | 1
Vaginal infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 2
Weight loss (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes